CLINICAL TRIAL: NCT00377442
Title: A Randomized, Open-label Crossover Study to Investigate the Potential Interaction Between GK Activator (2) and Simvastatin in Patients With Type 2 Diabetes
Brief Title: A Drug-Drug Interaction Study of GK Activator (2) and Simvastatin in Patients With Type 2 Diabetes.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NP20413
Record Dates: First submitted 2006-09-15; First posted 2006-09-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Simvastatin

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: GK Activator (2)
- 2 (Experimental)
  Interventions: Drug: Simvastatin
- 3 (Experimental)
  Interventions: Drug: GK Activator (2); Drug: Simvastatin

INTERVENTIONS:
Drug: GK Activator (2) — 100mg po
  Arms: 1; 3
Drug: Simvastatin — 80mg po
  Arms: 2; 3

SUMMARY:
This study will assess the potential pharmacokinetic interaction between GK Activator (2) and simvastatin, and the potential effect of simvastatin on the glucose-lowering effect of GK Activator (2) in patients with type 2 diabetes. Patients will be randomized to one of 6 treatment sequences to receive single doses of a)GK Activator (2) 100mg po, b)simvastatin 80mg po and c)GK Activator (2) 100mg + simvastatin 80mg po. Dosing will take place on study days 1, 8 and 15, and there will be a 7-14 day follow-up period after the last dose. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18-75 years;
* type 2 diabetes mellitus;
* untreated, or taken off anti-diabetic or statin therapy >=2 weeks before study start.

Exclusion Criteria:

* type 1 diabetes mellitus, or latent autoimmune diabetes in adults;
* diabetic neuropathy, retinopathy or nephropathy;
* patients treated with insulin or PPAR gamma agonist within 6 weeks of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2006-08; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
AUC0-inf of GK Activator (2) and simvastatin acid. | Days 1, 8 and 15
AUC0-6h of plasma glucose from pre-dose to 6h post-dose. | Days 1, 8 and 15

SECONDARY OUTCOMES:
AUC0-6h of GK Activator (2) and simvastatin acid | Days 1, 8 and 15
AUC0-inf of M4 and simvastatin; CL/F, Cmax, tmax, t1/2. | Days 1, 8 and 15
Cmin, tmin, Cmax, tmax, plasma glucose. | Days 1, 8 and 15
AEs, laboratory parameters. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- United States (2):
  - San Antonio, Texas
  - Tacoma, Washington